CLINICAL TRIAL: NCT00453635
Title: A Multicenter Randomized Phase II Study of First Line Treatment With Sequential Administration of Docetaxel, Carboplatin and Herceptin Versus the Administration of Vinorelbine and Herceptin Combination in HER-2 Positive Patients With Metastatic Breast Cancer
Brief Title: Study With Docetaxel, Carboplatin and Herceptin Versus Vinorelbine and Herceptin in HER-2 (+) Metastatic Breast Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor accrual
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: D. Mavrudis, Hellenic Oncology Research Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/03.08
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: Cancer; Breast cancer; First line treatment; Docetaxel; Carboplatin; Herceptin; Vinorelbine
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Docetaxel; Carboplatin; Trastuzumab; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Docetaxel + Carboplatin + Herceptin (D/Carbo/Her)
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Drug: Herceptin
- 2 (Experimental): Vinorelbine + Herceptin (VHer)
  Interventions: Drug: Herceptin; Drug: Vinorelbine

INTERVENTIONS:
Drug: Docetaxel — Docetaxel at the dose of 75mg/m^2 IV on day 1 every 3 weeks for 6 consecutive cycles
  Other Names: Taxotere
  Arms: 1
Drug: Carboplatin — Carboplatin at the dose of 5 AUC IV on day 1 every 3 weeks for 6 consecutive cycles
  Arms: 1
Drug: Herceptin — Herceptin 8 mg/Kg on day 1 for the first cycle and 6 mg/Kg for the 5 remaining cycles, IV, every 3 weeks
Drug: Vinorelbine — Vinorelbine at the dose of 60mg/m^2 per os,weekly
  Other Names: Navelbine
  Arms: 2

SUMMARY:
This trial will compare the efficacy of sequential administration of Docetaxel, Carboplatin and Herceptin versus the administration of Vinorelbine and Herceptin combination as first line treatment in HER-2 positive patients with metastatic breast cancer.

DETAILED DESCRIPTION:
Herceptin, a humanized monoclonal antibody directed against the extracellular domain of the transmembrane glycoprotein HER2/neu (c-erbB-2), is a valuable option in the treatment of women with HER2-positive metastatic breast cancer. The combination of Herceptin and chemotherapy yielded significantly better results than chemotherapy alone in response, time to progression, and survival time. Whether the combination of Docetaxel, Carboplatin and Herceptin versus the administration of Vinorelbine and Herceptin combination in HER-2 positive patients with metastatic breast cancer is preferable is not yet known.

ELIGIBILITY:
Inclusion Criteria:

* Performance status (WHO) 0-2
* Histologically confirmed metastatic breast adenocarcinoma (stage IV) without any prior chemotherapy received
* HER-2 overexpression 2+ or 3+ using IHC or FISH +
* Measurable disease not in a prior irradiation field (no other concurrent chemotherapy agents)
* No more than 25% of myeloproductive bone marrow irradiated (more than 4 weeks since prior radiotherapy and recovered)
* More than 6 months since prior adjuvant or neoadjuvant chemotherapy and recovered
* No prior first line chemotherapy for metastatic disease
* Endocrine therapy is allowed as adjuvant or first line treatment for metastatic disease
* Paraffin block from the primary tumor available in the research lab
* Adequate bone marrow function (absolute neutrophil count > 1000/mm^3, platelet count > 100000/mm^3, hemoglobin > 9 gr/mm^3)
* Adequate liver (Bilirubin < 1.5 times upper limit of normal and SGOT/SGPT < 2 times upper limit of normal) and renal function (creatinine < 2mg/dl)
* Adequate cardiac function (LVEF > 50%)
* Informed consent

Exclusion Criteria:

* Pregnant or nursing
* Concurrent agents ketoconazole, macrolide antibiotics, zidovudine which may induce P-450 cytochrome
* Positive pregnancy test
* Motor or sensory neuropathy > grade 1 according to NCIC Τoxicity Criteria
* Patients with brain metastatic disease who has not been irradiated or uncontrolled brain metastatic disease after irradiation
* History of allergic reaction attributed to docetaxel
* Psychiatric illness or social situation that would preclude study compliance
* Other concurrent uncontrolled illness.
* Other invasive malignancy within the past 5 years except cured basal cell skin carcinoma and cervical carcinoma in situ

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2003-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Time to progression between the two treatment arms | 1 year

SECONDARY OUTCOMES:
Overall survival | 1 year
Toxicity profile | During the time of chemotherpy

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Mavroudis, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (10):
- Greece (10):
  - University Hospital of Crete, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - Marika Iliadis" Hospital of Athens, Dep of Medical Oncology, Athens
  - State General Hospital of Larissa, Athens
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki